CLINICAL TRIAL: NCT03654859
Title: Silesian Registry of Out-of-Hospital Cardiac Arrests
Acronym: SIL-OHCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: Voivodeship Rescue Service in Katowice (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01012018
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2021-12

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: OHCA; cardiac arrest; cardiopulmonary resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cardiopulmonary resuscitation — no pre-specified

SUMMARY:
Silesian Registry of Out-of-Hospital Cardiac Arrests (SIL-OHCA) which is an initiative of the Voivodeship Rescue Service in Katowice in cooperation with the Silesian Center for Heart Diseases in Zabrze is a prospective, population-based registry of out-of-hospital cardiac arrests (OHCA). The main aim of the SIL-OHCA is to asses the frequency of OHCA in the population of Upper Silesia and analyze prognostic factors for long-term survival in patients with OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest treated by emergency medical services of Voivodeship Rescue Service in Katowice.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The area covered by the registry is a part of Silesian Voivodeship, Poland, which is the region of activity of Voivodeship Rescue Service in Katowice. There are 2,700,000 inhabitants in the area covered by the registry. All cases of out-of-hospital cardiac arrest with cardiopulmonary resuscitation started or continued by emergency medical services of Voivodeship Rescue Service in Katowice, as well as cases in which resuscitation is not attempted will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1560 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months

SECONDARY OUTCOMES:
30-day survival or survival to discharge | 30 days
Any return of spontaneous circulation | from OHCA until transfer to the hospital or decision to withdraw CPR (assessed up to 24 hours after OHCA)
  the occurence of any return of spontaneous circulation after cardiac arrest
Event survival | within first 24 hours after OHCA
  transfer to the hospital with sustained ROSC

CONTACTS AND LOCATIONS:
Locations (1):
- Voivodeship Rescue Service, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Undecided